CLINICAL TRIAL: NCT05055921
Title: A Clinical Feasibility Study to Evaluate the Safety and Performance of Low-Energy Therapy in Patients With Atrial Fibrillation (US)
Brief Title: MultiPulse Therapy (MPT) for AF (US)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor ceased operations
Sponsor: Cardialen, Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CL007 (US)
Record Dates: First submitted 2021-08-17; First posted 2021-09-24 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Multi-Pulse Therapy as delivered from the Cardialen External Stimulation System (CESS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Multi Pulse Therapy as delivered from the Cardialen External Stimulation System (Experimental): Subjects will have AF induced and the Cardialen External Stimulation System (CESS) device will deliver electrical stimulation to terminate the arrhythmia.
  Interventions: Device: Multi Pulse Therapy as delivered from the Cardialen External Stimulation System

INTERVENTIONS:
Device: Multi Pulse Therapy as delivered from the Cardialen External Stimulation System — The Cardialen External Stimulation System (CESS) is the research delivery system for the proprietary Cardialen MultiPulse Therapy (MPT). The CESS is a custom designed and built research device. It is comprised of off-the-shelf commercial components (power supplies, waveform generators, laptop computer, monitor, rack, ECG system, leads, etc.) combined with a custom electrical circuit board and custom software.
  Other Names:
  * Unpinning Termination Therapy
  * Multi-stage therapy
  * Multi-stage electrotherapy
  * MultiPulse Therapy

SUMMARY:
Assess the clinical safety and feasibility of MultiPulse Therapy (MPT) electrical stimulation waveform sequence in terminating paroxysmal and persistent atrial fibrillation.

DETAILED DESCRIPTION:
A prospective non-randomized feasibility study involving acute testing of MPT in subjects with paroxysmal and persistent AF during clinically indicated atrial fibrillation catheter ablation procedure.

Subjects will be split into 2 cohorts depending on status at time of procedure.

1. In Atrial Fibrillation at time of procedure (Clinical AF)
2. In Normal Sinus Rhythm at time of procedure

Subjects will be evaluated at the visits for the Clinically-Indicated Procedure per standard of care. A single follow-up at up to 30 days post-procedure is required to assess subjects for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 80 years of age
2. Willing and able to comply with the study protocol, provide a written informed consent
3. Currently indicated for atrial catheter ablation due to paroxysmal or early persistent atrial fibrillation
4. Current treatment and compliance with standard anticoagulation regimen, including uninterrupted OAC, with acceptable coagulation status, as determined by the Principal Investigator

Exclusion Criteria:

The subject must not meet any of the following exclusion criteria:

1. Life expectancy of 1 year or less
2. AF due to reversible causes (e.g., hyperthyroidism, valve disease)
3. History of DC Cardioversion which failed to convert to AF to Normal Sinus Rhythm
4. Currently in AF for more than 3 months continuously
5. Chronic, long-standing persistent, or permanent atrial fibrillation
6. Allergy or contraindication to anticoagulation therapy
7. Presence of intracardiac thrombus (confirmed with TEE or ICE)
8. Existing Left Atrial Appendage closure device
9. Severely Dilated Left Atrium >5cm
10. LVEF<35%
11. NYHA Class III or IV heart failure at the time of enrollment
12. History of embolic stroke, Transient Ischemic Attack (TIA) or other thromboembolic event within the preceding 3 months.
13. Known hyper-coagulable state that increases risk of thrombus
14. History of myocardial infarction or coronary revascularization within the preceding 3 months.
15. History of sustained ventricular arrhythmia or cardiac arrest
16. Presence of chronically implanted lead in the CS
17. Presence of ventricular assist device, including intra-aortic balloon pump
18. Documented bradycardia (<40 BPM) at the time of the study
19. Morbid obesity: BMI>39 kg/m2
20. Presence of any prosthetic cardiac valve
21. History of significant tricuspid valvular disease requiring surgery
22. Moderate to severe mitral valve regurgitation (>40% regurgitation fraction)
23. Cognitive or mental health status that would interfere with study participation and proper informed consent
24. Cardiovascular anatomical defects that would complicate placement of the stimulation leads required by the protocol, including congenital heart disease and cardiac vein anomalies per the Investigator's discretion
25. Pregnancy confirmed by test within 7 days of procedure.
26. Inability to pass catheters to heart due to vascular limitations
27. Cardiovascular surgery or intervention within 1 month prior to enrollment or planned for up to 1 month after enrollment (other than the planned treatment procedure)
28. Active endocarditis
29. Any other medical condition which may affect the outcome of this study or safety of the subject as determined by the investigator
30. History of hemodynamic compromise due to valvular heart disease
31. Unstable CAD as determined by the investigator
32. Severe proximal three-vessel or left main coronary artery disease without revascularization as determined by the investigator
33. History of Hypertrophic Cardiomyopathy, Arrhythmogenic Right Ventricular Dysplasia, Congenital Heart Anomaly, Cardiac Amyloidosis or Cardiac Sarcoidosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The safety of MPT for the treatment of atrial fibrillation in subjects | Acutely at the time of the study procedure
  Reported Adverse Events following MPT delivery
The safety of MPT for the treatment of atrial fibrillation in subjects | At 30 day post procedure
  Reported Adverse Events following MPT delivery
Enhanced ability of MPT to stop atrial fibrillation | Acutely following MPT delivery
  Compare voltages at which MPT successfully terminated AF against a previous Cardialen AF study (CL001 / NCT02257112)
Ability of MPT to stop atrial fibrillation | Acutely following MPT delivery
  Determine rate of conversion from AF to NSR

CONTACTS AND LOCATIONS:
Overall Officials: John D Hummel, MD, Principal Investigator — Ohio State University (OSU) Wexner Medical Center
Locations (2):
- United States (2):
  - Minneapolis Veterans Administration Hospital, Minneapolis, Minnesota
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janardhan AH, Gutbrod SR, Li W, Lang D, Schuessler RB, Efimov IR. Multistage electrotherapy delivered through chronically-implanted leads terminates atrial fibrillation with lower energy than a single biphasic shock. J Am Coll Cardiol. 2014 Jan 7-14;63(1):40-8. doi: 10.1016/j.jacc.2013.07.098. Epub 2013 Sep 26. PMID 24076284
- [Background] Li W, Janardhan AH, Fedorov VV, Sha Q, Schuessler RB, Efimov IR. Low-energy multistage atrial defibrillation therapy terminates atrial fibrillation with less energy than a single shock. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):917-25. doi: 10.1161/CIRCEP.111.965830. Epub 2011 Oct 6. PMID 21980076
- [Background] Efimov I, Ripplinger CM. Virtual electrode hypothesis of defibrillation. Heart Rhythm. 2006 Sep;3(9):1100-2. doi: 10.1016/j.hrthm.2006.03.005. Epub 2006 Mar 10. No abstract available. PMID 16945810
- [Background] Ambrosi CM, Ripplinger CM, Efimov IR, Fedorov VV. Termination of sustained atrial flutter and fibrillation using low-voltage multiple-shock therapy. Heart Rhythm. 2011 Jan;8(1):101-8. doi: 10.1016/j.hrthm.2010.10.018. Epub 2010 Oct 19. PMID 20969974